CLINICAL TRIAL: NCT01829659
Title: The ACS Ethnicity Platelet Function Study
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ACS Brilinta AZ
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AA Ticagrelor: African Americans who present with acute coronary syndrome (ACS) to the cath lab, and receive ticagrelor during their hospital stay.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor

SUMMARY:
This study is being done to assess the effects of the CTP inhibitor on the function of your platelets (cells within your blood that are involved in the formation of blood clots) and to assess whether you have responded to the ticagrelor well enough to prevent the formation of blood clots within the stent or site in which angioplasty was performed.

Recent studies have looked at how racial differences can affect platelet reactivity, the way blood clots. But these studies have not looked at the way different racial backgrounds can affect the way the blood forms clots. Minorities, such as African-Americans are underrepresented. Therefore, we are conducting this platelet reactivity study to better understand if there are differences in how this drug affects African-Americans from how they affect Caucasian patients undergoing percutaneous coronary intervention and receiving ticagrelor. These data will be compared to a historical control of Caucasian patients who underwent similar platelet function testing.

ELIGIBILITY:
Inclusion Criteria:

* Female (post menopausal or surgically sterile) and/or male aged 18 years or older
* Presenting with ACS fulfilling the following:

  1. Symptoms or new ECG changes (ST segment elevation or depression of at least 1 mm in 2 or more contiguous leads on EKG)
  2. Elevation of biomarkers (CK-MB ≥2 ULN or troponin ≥ ULN)
* Self-identified as African-American
* Treatment with 75-100mg ASA daily

Exclusion Criteria:

* Any indication (atrial fibrillation, mitral stenosis or prosthetic heart valve, PE, DVT) for antithrombotic treatment during study period.
* Fibrinolytic therapy within 48 hours before randomization
* Concomitant therapy with a drug having possible interaction with ticagrelor. (concomitant therapy with a strong cytochrome P-450 3A inhibitor or inducer)
* Increased bleeding risk including: recent (<30 days) GI bleeding, any history of intracranial, intraocular, retroperitoneal, or spinal bleeding, recent (<30 days of dosing) major trauma, sustained uncontrolled hypertension (systolic blood pressure [SBP]>180mmHg or diastolic blood pressure [DBP]>100mmHg), history of hemorrhagic disorders that can increase the risk of bleeding, platelet count less than 100,000 mm3 or hemoglobin <10 g/dL.
* Any history of hemorrhagic stroke.
* Contraindication or other reason that ASA or ticagrelor should not be administered (e.g., hypersensitivity, active bleeding, major surgery within 30 days of dosing).
* Severe renal failure (creatinine clearance <30mL/min or patient requires dialysis)
* History of moderate or severe hepatic impairment with aspartate amino transferace, alanine amino transferase or total bilirubin > 1.5 x upper limit of the reference range.
* Pregnant or lactating women.
* Patients receiving any glycoprotein IIb/IIIa inhibitors <8 hours before platelet reactivity testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty African American patients with documented acute coronary syndrome who agree to participate in this clinical study and who sign an informed consent will be enrolled.
  Race determination will be based on a patient's self-report, but patients enrolled in the trial must also report that all four of their grandparents were of the same race as theirs. Other races (Asian, Native American, etc) will be excluded from this study.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Ticagrelor Inhibition | 1-2 days
  The primary objective of the study is to assess ticagrelor's inhibition of platelet activity using 3 assays simultaneously: VerifyNow P2Y12 (PRU), vasodilator-stimulated phosphoprotein phosphorylation (VASP) and light transmission aggregometry (LTA) in African-American patients presenting with ACS.

SECONDARY OUTCOMES:
Follow-up Adverse Events | 30 days
  To evaluate the safety of ticagrelor treatment in African-American patients by assessment of adverse-events up to 30-day follow-up time point.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Medstar Washington Hospital Center, Washington D.C., District of Columbia, United States